CLINICAL TRIAL: NCT00407173
Title: An Open-Label, Single-Dose, Parallel Group Study to Evaluate the Effects of Age and Gender on the Pharmacokinetics, Safety, and Tolerability of HCV-796 Administered Orally to Healthy Subjects
Brief Title: Study to Evaluate the Effects of Age & Gender on PK, Safety & Tolerability of HCV-796 Administered to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: ViroPharma (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3173A1-112
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
MeSH Terms: interventions — HCV 796

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HCV-796 1000mg single dose
  Interventions: Drug: HCV-796

INTERVENTIONS:
Drug: HCV-796 — HCV-796 1000mg single dose

SUMMARY:
This study is an open-label, single-dose, parallel group study to evaluate the effects of age and gender on the pharmacokinetics, safety, and tolerability of HCV-796 administered orally to healthy subjects.

ELIGIBILITY:
Inclusion:

* Men or nonlactating and nonpregnant women, aged 18 to 45, and >65 years.
* Men must agree to practice barrier contraception for 12 weeks after the last test article administration.
* Estimated (calculated) creatinine clearance must be within the age-appropriate normal range.

Exclusion:

* History of seizures.
* History of rhabdomyolysis.
* History of thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of HCV-796 in healthy men and women of different ages. | 7 days

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single oral dose of HCV-796 in healthy men and women of different ages. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- United States (2):
  - Gainesville, Florida
  - Philadelphia, Pennsylvania